CLINICAL TRIAL: NCT00760097
Title: Adjunctive Transcranial Direct Current Stimulation for Cognition in Major Depression
Acronym: aTDCS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Ian A. Cook, M.D., Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: aTDCS in MDD
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AtCDS (Experimental): Transcranial direct stimulation
  Interventions: Device: Transcranial direct stimulation

INTERVENTIONS:
Device: Transcranial direct stimulation — sessions of 20 minutes each

SUMMARY:
People who have depression often have symptoms besides sad mood. Cognitive symptoms, such as poor memory, concentration, and decision making, are associated with disability in many spheres of life, and these symptoms often persist even when antidepressant treatment improves other symptoms (mood, energy, sleep, anxiety). Antidepressants alone fail to produce full remission for many patients, so it is important to study adjunctive treatments which can be added onto medication treatment and help restore cognitive function. The method of transcranial direct current stimulation (tDCS) has been shown by others to improve working memory and cognitive functions, and also to help with other symptoms of depression. tDCS involves passing a small, constant current between saline-moistened pads placed on the scalp. In this proposed study, 20 individuals with major depression who have cognitive difficulties despite taking antidepressants will participate. Over the course of a two-week period, each person will receive 5 sessions of either active tDCS or inactive treatments, in addition to their medication. Each session lasts for 20 minutes, and will be administered on alternating days (M-W-F). Assessments of depressive symptoms, cognitive function, and brain activity will be made prior to any sessions, after the first one, and after the fifth (final) session; brain function will be assessed by measuring the brain's electrical activity ("brain waves").

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS), also sometimes termed "DC polarization" or "brain polarization," is a non-invasive procedure that has been used successfully as a therapeutic intervention in a number of patient populations. tDCS involves the passing of very weak currents through an area of interest of the brain, by placing electrodes on the scalp at the appropriate locations. DC polarization has been shown to alter the amplitude of evoked potentials in the visual cortex (Antal et al., 2004), and cortical processing in the parietal lobe also can be modulated by tDCS (Rogalewski et al., 2004). From a more physiologically-relevant perspective, tDCS of the motor cortex has been shown to improve motor function in patients following stroke (Hummel and Cohen, 2005; Hummel et al., 2006; Boggio et al., 2006b) when applied to the prefrontal cortex. tDCS has been shown to improve working memory in healthy individuals (Fregni et al., 2005b), and in individuals with major depressive episode. In MDD it has more recently been shown to improve depression rating self-report scores (Fregni et al., 2006a) and cognitive performance (Fregni et al., 2006b). Performance on a executive function task (go/no-go) was also shown to be enhanced with tDCS in adults with MDD (Boggio et al., 2006a). tDCS has been evaluated in subjects with Parkinson's disease and found to have therapeutics benefit (compared with inactive treatment) on the Unified Parkinson's Disease Rating Scale and neuropsychological measures (reaction time, pegboard task) as well as motor evoked potentials (Fregni et al., 2006c).

Several recent studies have affirmed the safety of tDCS. Iyer and colleagues (2005) showed that, in a sample of 103 subjects, no one asked for the tDCS procedure to be stopped due to discomfort. Gandiga and colleagues (2006) compared sham to active tDCS and showed no differences in self-report ratings of discomfort. Nitsche and colleagues (2004) performed structural MRI scans on healthy individuals who underwent 1 hour exposures to tDCS; they found no evidence of structural change in the brain or alterations in blood-brain barrier permeability.

With regard to persistent challenges in the management of MDD, individuals with depression have shown cognitive deficits, particularly in working memory and other frontal lobe functions (Dunkin et al., 2000; Sweeney et al., 2000 Jaeger et al., 2006; Rose and Ebmeier 2006; Rose et al., 2006) and declarative memory (e.g., Beaden et al., 2006). By improving cognitive function in subjects with cognitive complaints that persist despite pharmacotherapy, it may be possible to improve the completeness of recovery from depression and reduce any functional disability (Jaeger et al., 2006).

There are no published reports yet of the effects of tDCS on brain function in subjects with MDD. Cordance is a quantitative electroencephalography (QEEG) measure which allows for non-invasive measurement of regional brain function (Leuchter et al., 1994a, 1994b, 1999; Cook et al., 1998). It is sensitive to changes in brain function in subjects who are responding to treatment for MDD (Cook and Leuchter 2001; Cook et al., 2002, 2005; Leuchter et al., 2002) and is being evaluated for use a a biomarker which predicts treatment outcome in MDD (NIMH Project R01MH069217, Cook PI). It is well suited to evaluating brain function in subjects with MDD during a clinical trial experiment.

Our hypotheses are

1. Subjects who are randomized to receive active tDCS treatments will show greater improvement in cognitive task performance than subjects who receive inactive treatments.
2. Subjects who are randomized to receive active tDCS treatments will show greater improvement in depression symptom severity scores than subjects who receive inactive treatments.
3. Subjects who are randomized to receive active tDCS treatments will show greater changes in prefrontal brain function, as assessed with quantitative EEG cordance, than subjects who receive inactive treatments.

ELIGIBILITY:
Inclusion Criteria:

* Subject age is 18 to 75 years old
* Subject meets the DSM-IV diagnosis of Major Depressive Disorder based on the MINI, with a current major depressive episode in partial remission
* Subject has been receiving treatment with an antidepressant medication for ≥ 3 months at a therapeutic dose. Therapeutic doses will be operationalized as those ranges noted by the drug manufacturers in their respective Package Inserts.
* Subject's score on the 17-item Hamilton Depression Rating Scale (Ham-D) is > 8 despite treatment with antidepressant medication(s).
* Subject has subjective cognitive complaints.

Exclusion Criteria:

* Subject is mentally or legally incapacitated, unable to give informed consent
* Subject suffering from a cognitive, bipolar, or psychotic disorder on the on the basis of a MINI interview; in situations where there is ambiguity about the origin of cognitive symptoms (i.e. depression with cognitive symptoms VS early dementia) subjects will not be enrolled.
* Subject meeting criteria for an Axis II diagnosis that would interfere with completion of the protocol
* Known drug dependency or substance abuse within the past six months
* Subject has had a course of ECT, Transcranial Magnetic Stimulation (TMS), or Vagus Nerve Stimulation (VNS) within the six months prior to enrollment
* Unstable medical illness, any history of seizures, brain surgery, skull fracture, significant head trauma, or previous abnormal EEG
* Ham-D score > 25 despite pharmacotherapy
* Subject is a UCLA student or staff member directly under instruction or employment of any of the investigators
* Subject has a medical illness which might be exacerbated by tDCS treatments (e.g. skin abrasions or infection of the scalp might be exacerbated by the placement of the saline-moistened electrode pads)
* Subject is using any of the following medications which interfere with EEG measures of brain function: Anticholinergics, Barbiturates, Benzodiazepines, Sedating Antihistamines (e.g. diphenhydramine (Benadryl) would be exclusionary, but not loratadine (Claritin)).
* Subject declines to give the study personnel permission to discuss their depression and participation in this study with their treating physician.
* Subject has had a suicide attempt or other self-injurious behavior in the past 6 months
* Subject has an implanted pacemaker
* Subject has red/green colorblindness (cannot distinguish red from green)
* Subject's intake urine test is positive for drugs of abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To test our hypotheses, assessments of cognition, mood, and brain activity will be performed on three occasions | 6 visits

SECONDARY OUTCOMES:
ADVERSE EVENT REPORTS Subjects will be asked about adverse events at the end of each treatment session | 6 visits

CONTACTS AND LOCATIONS:
Overall Officials: Ian Cook, Dr., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute for Neuroscience, Los Angeles, California, United States